CLINICAL TRIAL: NCT06473142
Title: CORRELATION BETWEEN SHOULDER DYSFUNCTION and FRONTAL PLANE POSTURE in SUBACROMIAL IMPINGEMENT SYNDROME
Brief Title: RELATION BETWEEN BODY POSTURE and SHOULDER DYSFUNCTION
Status: Recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Amr Saad Tawfik Soliman, DOCTOR, Cairo University
Other Study IDs: P.T.REC/012/005179
Record Dates: First submitted 2024-06-18; First posted 2024-06-25 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-08

CONDITIONS: Subacromial Impingement Syndrome; Frontal Plane Postural
MeSH Terms: conditions — Shoulder Impingement Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The purpose of this study will be to investigate if there is any correlation between shoulder dysfunction and the lateral alignment of the spine, scapular dyskinesia, pelvic tilting angle, Shoulder height angle, and trunk side bending (strength and mobility) in the frontal plane in patients with unilateral SIS.

DETAILED DESCRIPTION:
This study will be conducted to answer the following question:

Is there any correlation between shoulder dysfunction and the lateral alignment of the spine, scapular dyskinesia, pelvic tilting angle, Shoulder height angle, and trunk side bending (strength and mobility) in the frontal plane in patients with unilateral SIS?

This study will be limited to:

1. Thirty four (34) patients with unilateral SIS.
2. Male and female subjects will be included between 20 and 40 years of age .
3. Shoulder pain and disability level will be measured using the Arabic version of shoulder pain and disability index (SPADI).
4. Thoracolumbar lateral deviation will be measured using a scoliometer.
5. Scapular dyskinesia will be measured using lateral scapular slide test (LSST).
6. The pelvic tilting angle and shoulder height angle will be evaluated using Kinovea software.
7. Trunk side bending ROM will be evaluated using a bubble inclinometer .
8. Trunk side bending strength will be evaluated using a handheld dynamometer.

Assumptions:

It will be assumed that:

1. The instructions given to all individuals will be clear with satisfying explanations for all assessment methods.
2. All individuals will follow the instructions.

Hypotheses:

It will be hypothesized that:

1. There will be no significant correlation between pain score and measured variables in patients with unilateral SIS:

   1. lateral spinal deviation
   2. scapular dyskinesia
   3. pelvic tilting angle in the frontal plane
   4. shoulder height angle in the frontal plane
   5. ipsilateral trunk lateral side bending ROM
   6. contralateral trunk lateral side bending ROM
   7. ipsilateral trunk lateral side bending strength
   8. contralateral trunk lateral side bending strength
2. There will be no significant correlation between disability score and measured variables in patients with unilateral SIS:

   1. lateral spinal deviation
   2. scapular dyskinesia
   3. pelvic tilting angle in the frontal plane
   4. shoulder height angle in the frontal plane
   5. ipsilateral trunk lateral side bending ROM
   6. contralateral trunk lateral side bending ROM
   7. ipsilateral trunk lateral side bending strength
   8. contralateral trunk lateral side bending strength

ELIGIBILITY:
Inclusion Criteria:

1. Non-athletic patients of both sexes.
2. referred by an orthopedic surgeon with a diagnosis of unilateral SIS (Stage I, or II).
3. Patients aged between 20 to 40 years.
4. BMI between 18.5 to 29.9 kg/m2.
5. having four or more of the following findings:

   * Shoulder pain that is located either anteriorly or laterally to the acromion process
   * Pain worsening by shoulder flexion and/or abduction
   * A painful movement arc ranging from 60° to 120°
   * A palpably painful greater tuberosity of the humerus
   * The pain is replicated using the supraspinatus empty-can test, A positive Neer impingement sign, external rotation resistance test, and a positive Hawkins sign.

Exclusion Criteria:

1. Systematic illnesses
2. Pregnancy
3. Any degenerative disorder or disc lesion affection of the spine
4. A history of upper limb or spinal surgery
5. Previous upper limb or spinal fractures
6. Post-traumatic shoulder pain
7. History of shoulder instability (positive Sulcus sign, positive apprehension test, and history of shoulder dislocation)
8. Clinical signs of cervical radiculopathy (pain related to cervical movements)
9. Adhesive capsulitis
10. Tumors
11. Shoulder labral or cartilage lesions
12. Capsular or ligamentous tears or avulsions
13. any apparent deformity in the lower limbs including leg length discrepancy.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Thirty four (34) patients with unilateral SIS. Male and female subjects will be included between 20 and 40 years of age with a BMI between 18.5 to 29.9 kg/m2.
Sampling Method: Non-Probability Sample
Enrollment: 34 (Estimated)
Dates: Start 2024-08-19 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-10-15 (Estimated)

PRIMARY OUTCOMES:
Thoracolumbar lateral deviation | 2 MONTHES
  will be measured using a scoliometer
Scapular dyskinesia | 2 monthes
  will be measured using lateral scapular slide test (LSST)
The pelvic tilting angle and shoulder height angle | 2 monthes
  will be evaluated using Kinovea software
Trunk side bending ROM | 2 Monthes
  will be evaluated using a bubble inclinometer
Trunk side bending strength | 2 monthes
  will be evaluated using a handheld dynamometer
Shoulder pain and disability level | 2 monthes
  will be measured using the Arabic version of shoulder pain and disability index (SPADI)

CONTACTS AND LOCATIONS:
Locations (1):
- faculty of physical therapy Cairo university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
I do not have enough information right now

REFERENCES:
- [Background] Bhattacharyya R, Edwards K, Wallace AW. Does arthroscopic sub-acromial decompression really work for sub-acromial impingement syndrome: a cohort study. BMC Musculoskelet Disord. 2014 Sep 29;15:324. doi: 10.1186/1471-2474-15-324. PMID 25266967
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/